CLINICAL TRIAL: NCT01616173
Title: The Effects of Perineural Versus Intravenous Dexamethasone on Sciatic Nerve Blockade Outcomes
Brief Title: Analgesic Benefits of Perineural Versus Intravenous Dexamethasone in Patients Receiving Sciatic Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rohit Rahangdale, Assistant Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STU00058849
Record Dates: First submitted 2012-06-06; First posted 2012-06-11 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Fracture of Ankle
Keywords: Nerve Block; Anesthesia Recovery Period
MeSH Terms: conditions — Ankle Fractures | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perineural Dexamethasone (Active Comparator): Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine and perineural dexamethasone 8mg/2mL, and 50mL IV normal saline infusion
  Interventions: Drug: Dexamethasone
- Intravenous Dexamethasone (Active Comparator): Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine with saline and IV dexamethsone 8mg in 50mL infusion
  Interventions: Drug: Dexamethasone
- No Perioperative Steroids (Placebo Comparator): Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine with saline and 50mL infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — IV dexamethsone 8mg in 50mL (diluted in NS)
  Other Names: DECADRON
  Arms: Intravenous Dexamethasone
Drug: Dexamethasone — 8mg/2mL
  Other Names: DECADRON
  Arms: Perineural Dexamethasone
Drug: Saline — 2mL
  Other Names: Sodium chloride
  Arms: No Perioperative Steroids

SUMMARY:
Patients scheduled to have foot and ankle surgery will typically receive a single shot sciatic nerve block to serve as the primary anesthetic and as part of a multi-modal post-operative analgesic plan. The investigators are investigating the use of perineural dexamethasone together with local anesthetics can improve the quality of recovery for patients receiving sciatic nerve blocks for foot and ankle surgery.

DETAILED DESCRIPTION:
Patients scheduled to have foot and ankle surgery will typically receive a single shot sciatic nerve block to serve as the primary anesthetic and as part of a multi-modal post-operative analgesic plan. Perineural dexamethasone has been investigated as an adjuvant for brachial plexus nerve blocks but its effect on sciatic nerve block outcomes has yet to be determined. More importantly, it is not known whether the beneficial effect of perineural dexamethasone on analgesia duration leads to a better quality of surgical recovery. We hypothesized that perineural dexamethasone leads to a better quality of postsurgical recovery than intravenous dexamethasone or saline control.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients who are presenting for foot and ankle surgery and are candidates for a single injection sciatic nerve block to provide postoperative analgesia.
* Surgery confined to the foot and ankle.
* Patients aged 18-70 years.

Exclusion Criteria:

* ASA Classification of 4 or higher.
* Pre-existing neuropathy
* Coagulopathy
* Infection at the site
* Diabetes
* Non-English speaking or reading patients
* Systemic use of corticosteroids within 6 months of surgery
* Chronic opioid use
* Pregnancy
* Large (>3cm) skin incision around the medial aspect of the foot
* Any other contra-indication to regional anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Rahangdale, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Perineural Dexamethasone: Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine and perineural dexamethasone 8mg/2mL ,and 50mL IV normal saline infusion
- Intravenous Dexamethasone: Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine with saline/2mL and IV dexamethsone 8mg in 50mL infusion
- No Perioperative Steroids: Ultrasound guided sciatic nerve block with bupivicaine 0.5% with 1:300,000 epinephrine with saline/2mL and 50mL saline infusion
Period: Overall Study
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids
Started | 27 | 26 | 27
Completed | 27 | 24 | 27
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids | Total
Number analyzed (Participants) | 27 | 26 | 27 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [31 to 47] | 47 [32 to 55] | 39 [23 to 60] | 43 [30 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 11 | 37
  Male | 14 | 13 | 16 | 43

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery
Description: QoR-40 questionnaire instrument consists of 40 questions that examine 5 domains of patient recovery using a 5 point Likert scale: none of the time, some of the time, usually, most of the time and all of the time. The five domains include physical comfort, pain, physical independence, psychological support and emotional state. Global QoR-40 scores range from minimum of 40 to a maximum of 200. The scores are added together to compute a total score. A low score of 40 represents very poor quality of recovery while a high score, i.e. 200 represents outstanding quality of recovery.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids
Number analyzed (Participants) | 27 | 24 | 27
units on a scale | 181 [178 to 187] | 184 [181 to 188] | 181 [176 to 187]

2. Secondary Outcome: Opioid Consumption
Description: Postoperative opioid consumption was converted to equivalent dose of oral morphine at two weeks following surgery.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: mg/day
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids
Number analyzed (Participants) | 27 | 24 | 27
mg/day | 0 [0 to 7.5] | 0 [0 to 7] | 0 [0 to 7.5]

3. Secondary Outcome: Pain Scores
Description: Patients were asked to rate their pain score during activity on a 11-point scale (0 = no pain to 10 = excruciating pain).
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids
Number analyzed (Participants) | 27 | 24 | 27
units on a scale | 2 [0 to 4] | 2.5 [1 to 4] | 2 [0 to 5]

ADVERSE EVENTS:
Arm/Group | Perineural Dexamethasone | Intravenous Dexamethasone | No Perioperative Steroids
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/27

LIMITATIONS AND CAVEATS:
We enrolled a very specific surgical patient population and all surgical procedures required a saphenous nerve block and the pain in the saphenous nerve distribution could have affected some of our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes